CLINICAL TRIAL: NCT03665402
Title: Clinical Trial to Investigate the Appropriate Dose of Isoniazid According to NAT2 Polymorphism Status in Korean Subjects
Brief Title: A Pharamcogenomic Study for Isoniazid According to NAT2 Polymorphism Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INH NAT2
Record Dates: First submitted 2018-08-21; First posted 2018-09-11 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2018-12

CONDITIONS: Tuberculosis; Drug-Induced Liver Injury; Adverse Drug Event
MeSH Terms: conditions — Tuberculosis; Chemical and Drug Induced Liver Injury; Drug-Related Side Effects and Adverse Reactions | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rapid metabolizer (Standard treatment) (Active Comparator): Standard isoniazid dose regimen (300 mg qd)
  Interventions: Drug: Isoniazid
- Slow metabolizer (Standard treatment) (Active Comparator): Standard isoniazid dose regimen (300 mg qd)
  Interventions: Drug: Isoniazid
- Slow metabolizer (PGx treatment) (Experimental): Decreased isoniazid dose regimen (200 mg qd)
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Isoniazid — One of the first line anti-tubercolosis drug

SUMMARY:
A clinical trial to investigate the appropriate dose of isoniazid according to NAT2 polymorphism status in Korean subjects

ELIGIBILITY:
Inclusion Criteria:

* Agreement with written informed consent
* Adult healthy male or female subject age 20 to 45

Exclusion Criteria:

* Clinically significant, active gastrointestinal system, cardiovascular system, pulmonary system, renal system, endocrine system, blood system, digestive system, central nervous system, mental disease or malignancy
* Medication with any drug which may affect the pharmacokinetics of isoniazid within 14 days
* Previously donate whole blood within 30 days or Previously participated in other trial within 60 days
* Subject with known for hypersensitivity reactions to isoniazid
* Subject who can not perform contraception during study periods
* Female woman who are pregnant or are breast feeding
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-13 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Liver toxicity | up to 4 weeks
  Number of participants with drug-induced liver injury as assessed by below criteria.
  * AST or ALT > 5 ULN
  * AST or ALT > 3 ULN and total bilirubin > 2 ULN (Hy's law case)
  * ALT ratio/ALP ratio > 5

SECONDARY OUTCOMES:
Drug exposure | Day 1 and day 29 0, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 post-dose
  Plasma isoniazid concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No